CLINICAL TRIAL: NCT04896684
Title: Chronic Intestinal Pathologies Analytical Cohort at TouLouse
Acronym: CAPITOL
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/21/0038
Record Dates: First submitted 2021-05-03; First posted 2021-05-21 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Inflammatory Bowel Diseases; Colon Cancer
Keywords: Intestinal Bowel syndrome; Inflammatory Bowel Disease; colon cancer screening; data and biological collection
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colonic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — colon biopsies, blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient screened or followed-up for IBS or IBD or colorectal cancer: Blood and colon biopsy sampling
  Interventions: Biological: blood and intestinal biopsy sampling

INTERVENTIONS:
Biological: blood and intestinal biopsy sampling — 24 mL of blood and 10 intestinal biopsies will be sampled

SUMMARY:
In the general population, the percentage of people with at least one digestive disease is 16.7%. Among these digestive diseases, inflammatory bowel disease (IBD), irritable bowel syndrome (IBS) and patients who should benefit from digestive examinations as part of a screening oriented either by the patient's family history or following the performance of an immunological screening test ( FIT) in the stool will be studied. The aim of this project is to build a biological collection with associated clinical data for research projects.

DETAILED DESCRIPTION:
In the general population, the percentage of people with at least one digestive disease is 16.7%. Among these digestive diseases, two of them namely inflammatory bowel disease (IBD) and irritable bowel syndrome (IBS) will be more particularly studied. This interest is based on the increasing frequency of these two pathologies, their chronicities but above all the limited physiopathological data available. In addition, it seems interesting to study a third population, namely patients who should benefit from digestive examinations as part of a screening oriented either by the patient's family history or following the performance of an immunological screening test ( FIT) in the stool. The study of this population is part of an improvement in knowledge on the carcinogenesis of colorectal cancer.

To study these populations, blood, serum, plasma and tissues from colonous biopsies or surgical samples will be collected.

This cohort will make it possible to study, among other things, the pathophysiology of chronic diseases of the small intestine and the colon (IBD, IBS, screening) in order to improve their management through the development of new biomarkers and therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring endoscopic explorations for screening or follow-up in the context of a suspected IBS or IBD or colorectal cancer Or
* Patient with IBD requiring surgical management
* Patient over 18 years old
* Patient able to read and understand the information leaflet
* Patients who have given their consent to participate in the study
* Patients affiliated to a social security system (including AME)

Exclusion Criteria:

* Patients who have received antibiotic treatments in the 10 days preceding endoscopic exploration
* Pregnant or breastfeeding patients
* Patients under 18 years old
* Patients under guardianship or curatorship
* Patients unable to sign a free and informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Biological collection associated with clinical data | Baseline
  Set up a biological collection associated with clinical data on main intestinal tract diseases in order to understand their physiopathology
Biological collection associated with clinical data | pre-intervention/procedure/surgery
  Set up a biological collection associated with clinical data on main intestinal tract diseases in order to understand their physiopathology

SECONDARY OUTCOMES:
Identify new potential therapeutic molecules | Baseline
  Assessment of new treatment on organoids made thanks to intestinal biopsies
Optimize treatment success rates for IBD | Baseline
  Assessment of new treatment on organoids made thanks to intestinal biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Bournet, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Rangueil University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No